CLINICAL TRIAL: NCT02491892
Title: Open-Label, Phase II, Multicenter, Randomized Study of Efficacy and Safety for Two Different Doses of a Recombinant Humanized Antibody to HER2 (rhuMAb 2C4) Administered Every 3 Weeks to Patients With Metastatic Breast Cancer With Low Expression of HER2
Brief Title: A Study of Pertuzumab in Participants With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO16934
Record Dates: First submitted 2015-06-11; First posted 2015-07-08 (Estimated); Results first posted 2015-08-25 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab

ARMS (2):
- Pertuzumab 1050 mg (Experimental): Participants will not receive a loading dose, but will receive pertuzumab 1050 milligrams (mg) via intravenous (IV) infusion every 3 weeks until unacceptable toxicity or disease progression.
  Interventions: Drug: Pertuzumab
- Pertuzumab 420 mg (Experimental): Participants will receive a loading dose of 840 mg via IV infusion at the first infusion of pertuzumab, followed by a maintenance dose of 420 mg every 3 weeks until unacceptable toxicity or disease progression.
  Interventions: Drug: Pertuzumab

INTERVENTIONS:
Drug: Pertuzumab — Participants will receive one of two IV treatment regimens with pertuzumab: either 420 mg every 3 weeks, with an initial 840-mg loading dose, or 1050 mg every 3 weeks with no loading dose administered.
  Other Names: rhuMAb 2C4

SUMMARY:
This study will evaluate the efficacy and safety of pertuzumab (rhuMAb 2C4) in participants with metastatic breast cancer which has progressed during or after standard chemotherapy and which is not amenable to curative therapy. Those who are maintaining a response to therapy or who have stable disease at the end of the formal study period will continue treatment until disease progression or unacceptable toxicity. Approximately 120 participants will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Females at least 18 years of age
* Histologically-confirmed metastatic breast cancer with low HER2 expression and at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST)
* Karnofsky performance status at least 80%
* Disease progression on/after up to 2 different chemotherapy regimens, including an anthracycline-containing therapy
* Left ventricular ejection fraction (LVEF) at least 50%
* Adequate liver function

Exclusion Criteria:

* Pleural effusions, ascites, or bone lesions as the only manifestation(s) of cancer
* Pulmonary or central nervous system (CNS) metastases
* Chemotherapy, radiotherapy, or immunotherapy within 4 weeks; or hormone therapy within 2 weeks of Day 1
* Previous treatment with any drug that targets the HER2 receptor family
* Previous treatment with corticosteroids as cancer therapy
* History of significant cardiac disease
* Major surgery or trauma within 4 weeks of Day 1
* Pregnant or lactating women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2003-02; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (17):
- Australia (3):
  - Camperdown
  - Fitzroy
  - Geelong
- Namur, Belgium
- Finland (2):
  - Helsinki
  - Tampere
- Germany (3):
  - Hamburg
  - Herne
  - München
- Italy (2):
  - Milan
  - Parma
- Amsterdam, Netherlands
- Spain (2):
  - Barcelona
  - Valencia
- United Kingdom (3):
  - Edinburgh
  - London
  - Manchester

RESULTS

PARTICIPANT FLOW:
Groups:
- Pertuzumab 420 mg: Participants received a loading dose of 840 milligrams (mg) via intravenous (IV) infusion at the first infusion of pertuzumab, followed by a maintenance dose of 420 mg every 3 weeks until unacceptable toxicity or disease progression.
- Pertuzumab 1050 mg: Participants did not receive a loading dose, but received pertuzumab 1050 mg via IV infusion every 3 weeks until unacceptable toxicity or disease progression.
Period: Overall Study
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Started | 41 | 38
Treated | 41 | 37 (One participant was randomized but died before receiving study medication.)
Completed | 0 | 0
Not Completed | 41 | 38
Not completed — Adverse Event | 1 | 1
Not completed — Death | 1 | 1
Not completed — Lack of Efficacy | 37 | 36
Not completed — Refused Treatment | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: All randomized participants who received at least one dose of pertuzumab.
Groups:
- Pertuzumab 420 mg: Participants received a loading dose of 840 mg via IV infusion at the first infusion of pertuzumab, followed by a maintenance dose of 420 mg every 3 weeks until unacceptable toxicity or disease progression.
- Total: Total of all reporting groups
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg | Total
Number analyzed (Participants) | 41 | 37 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (10.04) | 53.5 (8.72) | 54.4 (9.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 37 | 78
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Best Overall Response of Confirmed Complete Response (CR) or Partial Response (PR)
Description: Objective tumor response was assessed using Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed CR was defined as the disappearance of all target lesions, and confirmed PR was defined as at least at 30 percent (%) decrease in the sum of the longest diameters of target lesions. Response was to be confirmed at follow-up assessment completed within 4 weeks of the first documented response. The percentage of participants achieving a best overall response of CR or PR was calculated as [number of participants meeting the above criteria divided by the number analyzed] multiplied by 100.
Time Frame: Up to approximately 1 year (at Baseline; every 6 weeks for the first 8 cycles, then every 12 weeks until progression or death; and up to 4 weeks after initial response)
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Number analyzed (Participants) | 41 | 37
percentage of participants | 4.9 | 0

2. Secondary Outcome: Time to Response Among Participants Achieving a Best Overall Response of Confirmed CR or PR
Description: Objective tumor response was assessed using RECIST. Confirmed CR was defined as the disappearance of all target lesions, and confirmed PR was defined as at least at 30% decrease in the sum of the longest diameters of target lesions. Response was to be confirmed at follow-up assessment completed within 4 weeks of the first documented response. Time to response was defined as the time from treatment start to first documented response (ie, CR or PR). Participants with stable disease (SD) were censored from the last tumor assessment, and those with progressive disease (PD) or death were assigned an artificial censoring time of 1000 days. Time to response was estimated using Kaplan-Meier and expressed in weeks.
Time Frame: as for outcome 1
Population: ITT Population.
Measure: Median (Full Range); unit: weeks
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Number analyzed (Participants) | 41 | 37
weeks | 12.1 [6.1 to 18.0] | NA [NA to NA] — Value could not be determined because no participants achieved CR or PR.

3. Secondary Outcome: Duration of Response Among Participants Achieving a Best Overall Response of Confirmed CR or PR
Description: Objective tumor response was assessed using RECIST. Confirmed CR was defined as the disappearance of all target lesions, and confirmed PR was defined as at least at 30% decrease in the sum of the longest diameters of target lesions. Response was to be confirmed at follow-up assessment completed within 4 weeks of the first documented response. Duration of response was defined as the time from first documented response (ie, CR or PR) to PD or death. Participants who did not experience PD or death were censored from the last tumor assessment. Duration of response was estimated using Kaplan-Meier and expressed in weeks.
Time Frame: as for outcome 1
Population: ITT Population.
Measure: Median (Full Range); unit: weeks
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Number analyzed (Participants) | 41 | 37
weeks | 24.6 [18.1 to 31.0] | NA [NA to NA] — Value could not be determined because no participants achieved CR or PR.

4. Secondary Outcome: Percentage of Participants Achieving a Best Overall Response of Confirmed CR
Description: Objective tumor response was assessed using RECIST. Confirmed CR was defined as the disappearance of all target lesions. Response was to be confirmed at follow-up assessment completed within 4 weeks of the first documented response. The percentage of participants achieving a best overall response of CR was calculated as [number of participants meeting the above criteria divided by the number analyzed] multiplied by 100.
Time Frame: as for outcome 1
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Number analyzed (Participants) | 41 | 37
percentage of participants | 0 | 0

5. Secondary Outcome: Duration of Response Among Participants Achieving a Best Overall Response of Confirmed CR
Description: Objective tumor response was assessed using RECIST. Confirmed CR was defined as the disappearance of all target lesions. Response was to be confirmed at follow-up assessment completed within 4 weeks of the first documented response. Duration of response was defined as the time from first documented response (ie, CR) to PD or death. Participants who did not experience PD or death were to be censored from the last tumor assessment. Duration of response was to be estimated using Kaplan-Meier.
Time Frame: as for outcome 1
Population: ITT Population.
Measure: Median (Full Range); unit: weeks
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Number analyzed (Participants) | 41 | 37
weeks | NA [NA to NA] — Value could not be determined because no participants achieved CR. | NA [NA to NA] — Value could not be determined because no participants achieved CR.

6. Secondary Outcome: Number of Participants Who Experienced PD or Death
Description: Objective tumor response was assessed using RECIST. PD was defined as the appearance of new lesion(s) or at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum obtained at Screening or during treatment. Participants who withdrew from the study early for insufficient therapeutic response without tumor assessment for PD were also included within the definition of PD.
Time Frame: as for outcome 1
Population: ITT Population.
Measure: Number; unit: participants
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Number analyzed (Participants) | 41 | 37
participants | 38 | 36

7. Secondary Outcome: Time to Progression
Description: Objective tumor response was assessed using RECIST. PD was defined as the appearance of new lesion(s) or at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum obtained at Screening or during treatment. Participants who withdrew from the study early for insufficient therapeutic response without tumor assessment for PD were also included within the definition of PD. Time to progression was defined as the time from treatment start to PD or death. Participants who did not experience PD or death were censored from the last tumor assessment. Time to progression was estimated using Kaplan-Meier and expressed in weeks.
Time Frame: as for outcome 1
Population: ITT Population.
Measure: Median (Full Range); unit: weeks
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Number analyzed (Participants) | 41 | 37
weeks | 6.1 [2.0 to 37.0] | 6.1 [2.7 to 36.3]

8. Secondary Outcome: Number of Participants Who Experienced PD or Withdrew From the Study Early
Description: Objective tumor response was assessed using RECIST. PD was defined as the appearance of new lesion(s) or at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum obtained at Screening or during treatment.
Time Frame: as for outcome 1
Population: ITT Population.
Measure: Number; unit: participants
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Number analyzed (Participants) | 41 | 37
participants | 41 | 37

9. Secondary Outcome: Time to Treatment Failure
Description: Objective tumor response was assessed using RECIST. PD was defined as the appearance of new lesion(s) or at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum obtained at Screening or during treatment. Time to treatment failure was defined as the time from treatment start to PD or early withdrawal from the study for death, toxicity, refusal/noncompliance, insufficient therapeutic response, or failure to return. Participants who did not experience PD or who did not withdraw from the study early were censored from the last tumor assessment. Time to treatment failure was estimated using Kaplan-Meier and expressed in weeks.
Time Frame: as for outcome 1
Population: ITT Population.
Measure: Median (Full Range); unit: weeks
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Number analyzed (Participants) | 41 | 37
weeks | 6.3 [2.0 to 80.1] | 6.0 [2.7 to 36.3]

10. Secondary Outcome: Percentage of Participants Who Died
Description: The percentage of participants who died was calculated as [number of participants with event divided by the number analyzed] multiplied by 100.
Time Frame: Up to approximately 2 years (from start of treatment until death)
Population: Safety Population: All randomized participants who received at least one dose of pertuzumab and had at least one post-baseline safety assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Number analyzed (Participants) | 41 | 37
percentage of participants | 46 | 32

11. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from treatment start to death. Participants who did not die during follow-up were to be censored from the last known alive date. Overall survival was to be estimated using Kaplan-Meier.
Time Frame: Up to approximately 2 years (from start of treatment until death)
Population: Median survival was not reached because the study program was terminated early. Analysis of the incomplete data set was not performed because it could potentially produce skewed or statistically irrelevant data.
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Percentage of Participants Achieving a Best Overall Response of SD
Description: Objective tumor response was assessed using RECIST. SD was defined as neither sufficient shrinkage to quality for PR nor sufficient increase to qualify for PD. The percentage of participants achieving a best overall response of SD was calculated as [number of participants meeting the above criteria divided by the number analyzed] multiplied by 100.
Time Frame: as for outcome 1
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Number analyzed (Participants) | 41 | 37
percentage of participants | 43.9 | 37.8

13. Secondary Outcome: Apparent Half-Life (t1/2) of Pertuzumab
Description: Serum samples were obtained for pharmacokinetic (PK) assessment using a receptor-binding, enzyme-linked immunosorbent assay (ELISA). Pertuzumab concentrations at each collection point were used to determine the apparent t1/2 by non-compartmental analysis, defined as the time elapsed for pertuzumab concentrations to decrease by 50%. The derived value was averaged among all participants and expressed in days.
Time Frame: Pre-dose and within 15 minutes of the end of infusion on Day 1 of each cycle, and on Days 8 and 15 of Cycles 1 and 2
Population: ITT Population. Participants with missing PK data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Number analyzed (Participants) | 38 | 36
days | 12.2 (3.9) | 11.4 (4.1)

14. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Pertuzumab
Description: Serum samples were obtained for PK assessment using a receptor-binding ELISA. The maximum observed pertuzumab concentration across all collection points was documented. Cmax was averaged among all participants and expressed in micrograms per milliliter (mcg/mL).
Time Frame: Pre-dose and within 15 minutes of the end of infusion on Day 1 of each cycle, and on Days 8 and 15 of Cycles 1 and 2
Population: ITT Population. Participants with missing PK data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Number analyzed (Participants) | 40 | 37
mcg/mL | 289 (107) | 409 (159)

15. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Pertuzumab
Description: Serum samples were obtained for PK assessment using a receptor-binding ELISA. The time of maximum observed pertuzumab concentration across all collection points was documented. Tmax was averaged among all participants and expressed in days.
Time Frame: Pre-dose and within 15 minutes of the end of infusion on Day 1 of each cycle, and on Days 8 and 15 of Cycles 1 and 2
Population: ITT Population. Participants with missing PK data were excluded from the analysis.
Measure: Median (Full Range); unit: days
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Number analyzed (Participants) | 40 | 37
days | 0.073 [0.052 to 7] | 0.073 [0.059 to 0.122]

16. Secondary Outcome: Area Under the Concentration-Time Curve (AUC) of Pertuzumab
Description: Serum samples were obtained for PK assessment using a receptor-binding ELISA. Pertuzumab concentrations at each collection point were used to determine AUC to the last measurable observation (AUClast) and AUC extrapolated to infinity (AUCinf) by non-compartmental analysis. The derived values were averaged among all participants and expressed in days by micrograms per milliliter (days*mcg/mL).
Time Frame: Pre-dose and within 15 minutes of the end of infusion on Day 1 of each cycle, and on Days 8 and 15 of Cycles 1 and 2
Population: ITT Population. Participants with missing PK data were excluded from the analysis, and the number of participants analyzed (n) is presented here.
Measure: Mean (Standard Deviation); unit: days*mcg/mL
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Number analyzed (Participants) | 40 | 37
days*mcg/mL
  AUClast (n=40,37) | 2517 (896) | 3465 (1051)
  AUCinf (n=38,36) | 3598 (1402) | 4750 (1527)

17. Secondary Outcome: Systemic Clearance (CL) of Pertuzumab
Description: Serum samples were obtained for PK assessment using a receptor-binding ELISA. Pertuzumab concentrations at each collection point were used to determine CL by non-compartmental analysis, defined as the rate at which pertuzumab was removed from the body. The derived value was averaged among all participants and expressed in milliliters per day (mL/day).
Time Frame: Pre-dose and within 15 minutes of the end of infusion on Day 1 of each cycle, and on Days 8 and 15 of Cycles 1 and 2
Population: ITT Population. Participants with missing PK data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Number analyzed (Participants) | 38 | 36
mL/day | 270 (113) | 247 (90)

18. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Pertuzumab
Description: Serum samples were obtained for PK assessment using a receptor-binding ELISA. Pertuzumab concentrations at each collection point were used to determine the Vss by non-compartmental analysis, defined as the theoretical volume at which the total amount of pertuzumab would be uniformly distributed to produce the desired concentration. The derived value was averaged among all participants and expressed in milliliters (mL).
Time Frame: Pre-dose and within 15 minutes of the end of infusion on Day 1 of each cycle, and on Days 8 and 15 of Cycles 1 and 2
Population: ITT Population. Participants with missing PK data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Number analyzed (Participants) | 38 | 36
mL | 4122 (1666) | 3527 (1369)

19. Secondary Outcome: Mean Residence Time (MRT) of Pertuzumab
Description: Serum samples were obtained for PK assessment using a receptor-binding ELISA. Pertuzumab concentrations at each collection point were used to determine the MRT by non-compartmental analysis. The derived value was averaged among all participants and expressed in days.
Time Frame: Pre-dose and within 15 minutes of the end of infusion on Day 1 of each cycle, and on Days 8 and 15 of Cycles 1 and 2
Population: ITT Population. Participants with missing PK data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Number analyzed (Participants) | 38 | 36
days | 16 (5) | 15 (6)

20. Secondary Outcome: Number of Participants Experiencing a Drop in Left Ventricular Ejection Fraction (LVEF) to a Value of Less Than 50%
Description: Echocardiography was performed to determine LVEF, defined as the volume of blood pumped from the left ventricle as a percentage of end-diastolic volume. Theoretically, LVEF may range from 0 to 100%. The number of participants experiencing a drop in LVEF greater than or equal to (≥) 10 or 15 percentage points to a final LVEF of less than (<) 50% is reported here.
Time Frame: Up to approximately 1 year (at Baseline; at the end of Cycles 2, 4, 8, 12, and 16; and up to 7 weeks following the last infusion)
Population: Safety Population.
Measure: Number; unit: participants
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Number analyzed (Participants) | 41 | 37
participants
  Drop ≥10 percentage points | 3 | 5
  Drop ≥15 percentage points | 3 | 3

ADVERSE EVENTS:
Time Frame: Up to approximately 1 year (from start of treatment until up to 7 weeks following the last infusion)
Arm/Group | Pertuzumab 420 mg | Pertuzumab 1050 mg
Serious Adverse Events (participants affected / at risk) | 10/41 | 8/37
Other Adverse Events (participants affected / at risk) | 36/41 | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pertuzumab 420 mg (N=41) | Pertuzumab 1050 mg (N=37)
Ascites (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Ejection fraction decreased (Investigations) | 2 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pertuzumab 420 mg (N=41) | Pertuzumab 1050 mg (N=37)
Diarrhoea (Gastrointestinal disorders) | 24 | 22
Nausea (Gastrointestinal disorders) | 12 | 13
Asthenia (General disorders) | 10 | 9
Vomiting (Gastrointestinal disorders) | 10 | 8
Abdominal pain upper (Gastrointestinal disorders) | 6 | 6
Anorexia (Metabolism and nutrition disorders) | 4 | 8
Headache (Nervous system disorders) | 7 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Fatigue (General disorders) | 5 | 5
Rash (Skin and subcutaneous tissue disorders) | 6 | 4
Stomatitis (Gastrointestinal disorders) | 4 | 4
Anaemia (Blood and lymphatic system disorders) | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Chest pain (General disorders) | 2 | 5
Dyspepsia (Gastrointestinal disorders) | 3 | 3
Ejection fraction decreased (Investigations) | 3 | 3
Mucosal inflammation (General disorders) | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 1
Paraesthesia (Nervous system disorders) | 3 | 2
Dizziness (Nervous system disorders) | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2
Urinary tract infection (Infections and infestations) | 2 | 2
Dysgeusia (Nervous system disorders) | 0 | 3
Dysuria (Renal and urinary disorders) | 1 | 2
Herpes simplex (Infections and infestations) | 1 | 2
Insomnia (Psychiatric disorders) | 0 | 3
Oesophagitis (Gastrointestinal disorders) | 1 | 2
Pyrexia (General disorders) | 3 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 2
Ear infection (Infections and infestations) | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 2

LIMITATIONS AND CAVEATS:
Recruitment was halted within the planned study design. The study was designed to stop recruitment following the interim analysis if the response rate (CR or PR) was <1 of 23 participants per arm after all participants completed at least 2 cycles.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.